CLINICAL TRIAL: NCT04465968
Title: Efficacy and Safety of Durvalumab Before and After Operation or Durvalumab as Maintenance Therapy After Chemoradiotherapy Against Superior Sulcus Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of CRT, Durvalumab and Surgery for SST
Acronym: DEEP_OCEAN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: AstraZeneca (Industry); Japan Agency for Medical Research and Development (Other Government); Japan Clinical Oncology Group (Other)
Responsible Party: Principal Investigator, Masahiro Tsuboi, MD, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1807C
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Superior Sulcus Tumor; Non-small Cell Lung Cancer Stage IIB; Non Small Cell Lung Cancer Stage III
Keywords: Superior Sulcus Tumor; Pancoast Tumor; Non-Small Cell Lung Cancer; Durvalumab; Multi-modality therapy; Neoadjuvant therapy
MeSH Terms: conditions — Pancoast Syndrome; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; S 1 (combination); durvalumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT + Durvalumab ± Surgery + Durvalumab (Experimental): Concurrent chemoradiotherapy (cisplatin+S-1+radiotherapy 66Gy)+2 courses of durvalumab followed by Surgery and adjuvant durvalumab for resectable SST or chemoradiotherapy (cisplatin+S-1+radiotherapy 66Gy) followed by maintenance durvalumab for unresectable SST.
  Interventions: Drug: Cisplatin; Drug: S1; Radiation: concurrent radiotherapy; Drug: Durvalumab; Procedure: Surgery

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60 mg/m2, IV, day 1
Drug: S1 — 80 - 120 mg/day, PO, day 1-14
Radiation: concurrent radiotherapy — 66 Gy/33 Fr
Drug: Durvalumab — preoperative durvalumab therapy within 28 days after chemoradiotherapy. Two courses are given every two weeks.
Procedure: Surgery — Surgery will be performed between day 15 and day 42 of the second course of preoperative durvalumab therapy after confirming that all surgical operation criteria are met.
Drug: Durvalumab — (For resectable SST) Postoperative durvalumab therapy will be started between day 28 and day 63 with the day of surgery as Day 1. Twenty-two courses are given as a 2-week course.
  Drug: Durvalumab 10 mg/kg/body, IV, day 1 (For unreectable SST) Additional durvalumab therapy between day 15 and day 28 of the second course of preoperative durvalumab therapy.
  Twenty-two courses are given as 2-week course. Drug: Durvalumab 10 mg/kg/body, IV, day 1

SUMMARY:
The safety and efficacy of multimodality treatment of pre- and post-operative durvalumab therapy after pre-operative chemoradiotherapy for resectable superior sulcus tumor (SST) and durvalumab maintenance therapy after chemoradiotherapy for unresectable SST

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of multimodality treatment of pre- and post-operative durvalumab therapy after pre-operative chemoradiotherapy for resectable superior sulcus tumor (SST) and durvalumab maintenance therapy after chemoradiotherapy for unresectable SST

ELIGIBILITY:
Inclusion Criteria:

1. A definite diagnosis of non-small cell lung cancer has been obtained by biopsy from the primary lesion.
2. Meet all of the following (UICC-TNM classification 8th edition). I. Regarding the primary lesion, meet one of the following on chest CT. i. Direct invasion of the chest wall at or above the height of the first rib (at least invasion of the parietal pleura) ii. Direct invasion of the subclavian artery or vein II. Regarding regional lymph nodes, meet either of the following by chest CT and FDG-PET/CT. Metastasis is also considered if lymph node metastasis is determined by either chest CT or FDG-PET/CT.

   i. cN0 ii. cN1 and no metastases to #10, #11, and #12 lymph nodes iii. cN3 (ipsilateral supraclavicular lymph node metastasis) and no metastases in regional lymph nodes (N1 and N2) other than "#13, #14 lymph nodes" III. No distant metastases (including intrapulmonary metastases in the same ling lobe and in a different lung lobe on the same side) on imaging tests including FDG-PET/CT
3. It is judged that radical resection is possible by lobectomy (including bilobectomy for 2 lobes), which satisfies the following [1] and [2].

   I. The board respiratory surgeon judges that none of the following is true based on the image findings.

   i. There is vertebral body infiltration that requires total spondylectomy ii. Presence of spinal cord infiltration iii. Invaded trachea or tracheal bifurcation iv. Invasion of aortic arch or ascending aorta v. Invading brachial plexus at C8 or higher vi. Esophageal infiltration that requires esophageal reconstruction for resection vii. Pneumonectomy is required for radical resection II. Meet all of the following. i. Predicted postoperative forced expiratory volume of 1 second (FEV1.0) ≥ 800 mL within 56 days before registration ii. SpO2 > 93% (room air) with the latest inspection value within 14 days before registration
4. Consult with the radiotherapy doctor and it is judged that all of the following are met.

   I. Radiation therapy is possible according to the protocol II. The irradiation field does not reach the hilum
5. The age of the registration date is 20 years or older and 75 years or yonger.
6. Performance status (PS) is 0 or 1 according to ECOG standards (PS must be described in medical records)
7. The presence or absence of measurable lesions is not required.
8. No history of following surgery irrespective of whether for a benign or malignant lesion.

   I. Thoracoscopic surgery or thoracotomy with excision of the affected lung or esophagus or mediastinum (however, a history of thoracoscopic surgery without wedge resection or lung, esophagus, or mediastinal resection (eg, pleural biopsy)) is allowed) II. Median sternotomy surgery (with or without organ resection) III. Pulmonary resection other than wedge resection of the contralateral lung (whether open-heart surgery or thoracoscopic surgery)
9. There is no history of chemotherapy, including treatment for other cancer types (including molecular targeted therapies and immune checkpoint inhibitors). However, the history of drug therapy as adjuvant therapy is allowed if it was completed more than 3 years ago. In addition, a history of hormone therapy for other cancer types is allowed.
10. If there is a history of radiotherapy including other cancer types, the lung, hilum, mediastinum, and supraclavicular fossa are not included in the irradiation field.
11. Chest CT does not show interstitial pneumonia or pulmonary fibrosis.
12. No history of complication of autoimmune disease or chronic or recurrent autoimmune disease. However, patients with type 1 diabetes which is well controlled by appropriate treatment, hyperthyroidism/hypothyroidism that requires only antithyroid drug/hormone replacement therapy, autoimmune skin disease that does not require systemic treatment (Pemphigus, psoriasis vulgaris, pemphigus vulgaris, vitiligo), and celiac disease controlled only by dietary control are regarded as eligible if they have been inactive in the past 5 years, even with a history of autoimmune complications or history.
13. No surgical treatment with general anesthesia within 14 days (2 weeks) before registration.
14. No systemic administration of steroids, other immunosuppressive drugs, or immunoglobulins within 28 days (4 weeks) before registration. However, those that meet the following conditions are allowed.

    I. Intranasal/inhalation/topical steroid injection or local steroid injection (for example, intra-articular injection) II. Systemic administration of steroid drugs at a dose of 10 mg/day or less in terms of prednisolone III. Steroids as premedication (eg CT premedication)
15. Can be taken orally.
16. No ischemic changes were observed on the latest 12-lead ECG within 28 days before registration. However, if a 12-lead electrocardiogram shows ischemic changes, echocardiography, exercise electrocardiography, etc. should be performed, and if it is judged that new treatment for ischemic heart disease is not necessary, it is qualified.
17. The latest inspection value within 14 days before registration (possible on the same day two weeks before the registration date) satisfies all of the following.

    I. White blood cell count ≧4,000/mm3 II. Hemoglobin ≥ 11.0 g/dL (no blood transfusion within 14 days before the blood sampling date of the test used for registration) III. Platelet count ≧10×104 /mm3 IV. Total bilirubin ≤ 2.0 mg/dL V. AST ≤ 75 U/L VI. ALT ≤ 75 U/L VII. Serum creatinine ≤ 1.2 mg/dL
18. Written informed consent from the patient to participate in the study.
19. The attending physician can judge that the enrolled patients understand the treatment and evaluation schedule of this study and can comply with them.

Exclusion Criteria:

1. Having active double cancer (simultaneous double cancer/multiple cancer and metachronous double cancer/multiple cancer with a disease-free period of 3 years or less, even if the disease-free period is less than 3 years, clinical The 5-year relative survival rate is similar to that of stage I prostate cancer, clinical stage 0 completely responded to radiation therapy, stage I laryngeal cancer, and complete excision of the following pathological stage cancers. History of cancer equivalent to 95% or more is not included in active double cancer/multiple cancer). Gastric cancer "adenocarcinoma (general type)": Stage 0-I, colon cancer (adenocarcinoma): Stage 0-I, rectal cancer (adenocarcinoma): Stage 0-I, esophageal cancer (squamous cell carcinoma, glandular) Squamous cell carcinoma, basal cell carcinoma): Stage 0, breast cancer (non-invasive ductal carcinoma, lobular carcinoma): Stage 0, breast cancer (invasive ductal carcinoma, lobular invasive carcinoma, Paget's disease): 0 Stage-IIA, endometrial cancer (endometrioid adenocarcinoma, mucinous adenocarcinoma): Stage I, prostate cancer (adenocarcinoma): Stage I-II, cervical cancer (squamous cell carcinoma): Stage 0, thyroid cancer (Papillary cancer, follicular cancer): stage I, stage II, stage III, renal cancer (clear cell carcinoma, chromophobe cell carcinoma): stage I, non-melanoma skin cancer, malignant melanoma without a definite diagnosis, etc. Lesions of intramucosal cancer
2. Has an infectious disease that requires systemic treatment (including active pulmonary tuberculosis).
3. When registering, a fever of 38.0°C or higher is generated.
4. Women who are pregnant, possibly pregnant, within 28 days of delivery, or breastfeeding. A man who wants a partner to become pregnant. Or a reproductive male or female patient who is not willing to use an effective contraceptive by Week 13 (Day 91) after the last dose of durvalumab (see 6.4.7.).
5. Participation in the study is considered to be difficult due to the combination of mental illnesses or symptoms that impair daily life.
6. Continuous systemic administration (oral or intravenous) of steroid drugs or other immunosuppressive drugs in excess of 10 mg/day in terms of prednisolone.
7. With uncontrolled diabetes.
8. With uncontrolled hypertension.
9. A gastrointestinal disorder accompanied by uncontrolled diarrhea.
10. With unstable angina (angina with onset or exacerbation of attack within the last 3 weeks) or a history of myocardial infarction within 6 months.
11. Poor valvular heart disease, dilated cardiomyopathy, hypertrophic cardiomyopathy, congestive heart failure, and arrhythmia.
12. Chest CT reveals severe emphysema.
13. Either HBs antigen, HCV antibody, or HIV1/2 antibody is positive.
14. Continuous use of flucytosine (Ancotil®) is required.
15. Participating in another clinical trial (excluding observational studies) during the 6 months prior to enrollment.
16. A history of allogeneic organ transplant.
17. A history of active primary immunodeficiency.
18. Live vaccines (BCG, polio, measles-rubella mixture, measles, rubella, mumps, chickenpox, yellow fever, rotavirus, etc.) have been administered within 30 days before registration.
19. Has hypersensitivity or allergy to the test drug or its additives used in this test.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival rate (3y-OS) | 3 years
  3-year overall survival rate

SECONDARY OUTCOMES:
3-year progression-free survival rate (3y-PFS) | 3 years
  3-year progression-free survival rate
5-year progression-free survival rate (5y-PFS) | 5 years
  5-year progression-free survival rate
5-year overall survival rate (5y-OS) | 5 years
  5-year overall survival rate
Mode of recurrence | 5 years
  Mode of recurrence in surgical cases
Local recurrence rate | 5 years
  Proportion of local failure in surgical cases
Objective response rate (ORR) | 1 year 6 months
  Objective response rate according to RECIST and iRECIST
Resection rate | 1 year 6 months
  Proportion of surgical cases
Pathological complete resection rate (R0 rate) | 1 year 6 months
  Proportion of pathologcal complete resection in surgical cases
Pathological complete response rate (pCR rate) | 1 year 6 months
  Proportion of pathologcal complete response in surgical cases
Major pathological response rate (MPR rate) | 1 year 6 months
  Determination of major pathologic response rate is based on the method by Hellmann et al. on the pathological section. The percentage of residual tumor cells is calculated as viable tumor cells / tumor area × 100 (%). Tumor area includes viable tumor cells and interstitial tissue such as fibrosis, necrosis, and inflammatory cells.
Operation time | 1 year 6 months
  Operation time in surgical cases
Blood loss | 1 year 6 months
  Intraoperative blood loss in surgical cases
Adverse event rate | 1 year 6 months
Incidences of serious adverse events | 1 year 6 months
Incidences of adverse events | 1 year 6 months

IPD SHARING:
Plan to Share IPD: No